CLINICAL TRIAL: NCT02557763
Title: Study of Oxford Unicompartmental Knee Arthroplasty to Determine Anterior Knee Pain, Pain Score, Knee Score and Functional Score Between Patients Without Severe Patellofemoral Arthritis and Patients With Severe Patellofemoral Arthritis
Brief Title: To Compare Anterior Knee Pain Between Non Severe and Severe Patellofemoral Arthritis After Oxford UKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonchana Pongcharoen, Associate Professor, Thammasat University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-EC-OT-0-091/57
Record Dates: First submitted 2015-05-07; First posted 2015-09-23 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
Keywords: Oxford UKA; anterior knee pain; lateral facet of patella
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Severe PF arthritis (Experimental): Oxford unicompartmental knee arthroplasty is partial knee replacement. Oxford unicompartmental knee arthroplasty is applied for medial compartmental of knee.
  Interventions: Device: Oxford unicompartmental knee arthroplasty
- non severe PF arthritis (Experimental): Oxford unicompartmental knee arthroplasty is partial knee replacement. Oxford unicompartmental knee arthroplasty is applied for medial compartmental of knee.
  Interventions: Device: Oxford unicompartmental knee arthroplasty

INTERVENTIONS:
Device: Oxford unicompartmental knee arthroplasty — The patients with medial osteoarthritis knee with patellofemoral arthritis were performed surgery and applied Oxford unicompartmental knee arthroplasty.
  Other Names: Oxford UKA

SUMMARY:
The aims of this study is to compare the results between patients without severe patellofemoral arthritis and patients with severe patellofemoral arthritis after mobile bearing UKA.

The investigators prospective compute the results including anterior knee pain, knee society score, pain score, functional score, range of motion, operative time, blood loss, and component alignment.

DETAILED DESCRIPTION:
The patients were performed surgery. The Oxford UKA was applied for all patient.

ELIGIBILITY:
Inclusion Criteria:

* anteromedial osteoarthritis knee,
* older than 40 years old,
* range of motion > 90 degrees,
* varus deformity < 25degrees,
* flexion contracture< 20degrees,
* intact anterior cruciate ligament

Exclusion Criteria:

* younger than 40,
* osteonecrosis of knee,
* rheumatoid,
* posttraumatic arthritis,
* absent of anterior cruciate ligament

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
visual analog scale for anterior knee pain | 1 year
  The 10-point visual analog scale is 0 representing no pain and 10 representing maximum pain experience.

SECONDARY OUTCOMES:
Knee society score | 1year
  The standard clinical evaluation system for reporting results for patients undergoing unicompartmental knee arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Boonchana Pongcharoen, MD, Principal Investigator — Thammasat University
Locations (1):
- Boonchana Pongcharoen, Pathum Thani, Changwat Pathum Thani, Thailand